CLINICAL TRIAL: NCT06724991
Title: Efficacy of Lower-Dose Versus Conventional-Dose of Insulin and Dextrose for Treatment of Mild and Moderate Hyperkalaemia in Emergency Department: a Randomised, Triple-Blinded, Non-Inferiority Trial
Brief Title: Lower Vs. Standard Insulin-Dextrose Doses for Treating Mild to Moderate Hyperkalemia in the Emergency Department
Acronym: IDK+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Khadijah Poh Yuen Yoong, Consultant Emergency Physician, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024101-14273; RSCH ID-24-06414-1Q3 (Other: National Medical Research Registry)
Record Dates: First submitted 2024-12-06; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hyperkalemia
Keywords: hyperkalemia; hypoglycemia; lower dose insulin; extravasation injury
MeSH Terms: conditions — Hyperkalemia; Hypoglycemia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Dose Therapy (Active Comparator): Traditional treatment involves a higher insulin dose with dextrose to mitigate hypoglycemia risk while effectively lowering potassium. Ingredients: Actrapid insulin, Dextrose 50% Dosage: 10 units of Actrapid insulin with 50 cc of Dextrose 50% Route of Administration: Intravenous (IV) Frequency: Administered as a single dose at the start of treatment Procedure: The conventional dose has been the standard of care but carries a significant risk of hypoglycemia.
  Interventions: Procedure: Conventional Dose Therapy
- Lower Dose Therapy (Experimental): Standard treatment of hyperkalemia includes insulin to shift potassium intracellularly and dextrose to mitigate the risk of hypoglycemia. This arm will be active intervention which means to compare with traditional dose of insulin and investigate if lower dose of insulin is non inferior in reducing serum potassium level in patient with mild and moderate hyperkalemia. Ingredients: Actrapid insulin, Dextrose 50% Dosage: 5 units of Actrapid insulin with 25 cc of Dextrose 50% Route of Administration: Intravenous (IV) Frequency: Administered as a single dose at the start of treatment Procedure: Lower-dose insulin is administered with dextrose to potentially reduce hypoglycemic risk while achieving effective potassium reduction.
  Interventions: Procedure: Lower Dose Therapy

INTERVENTIONS:
Procedure: Lower Dose Therapy — The group receiving the lower-dose therapy consists of 5 units of Actrapid (insulin) with 25cc of Dextrose 50%. This intervention is the focus of the clinical trial and is being investigated to determine if it achieves a comparable reduction in potassium levels with fewer potential complications. The aim is to establish it as a non-inferior alternative to conventional-dose therapy in the management of mild and moderate hyperkalemia.
  Arms: Lower Dose Therapy
Procedure: Conventional Dose Therapy — The group receiving the conventional-dose therapy, consisting of 10 units of Actrapid (insulin) with 50cc of Dextrose 50%, which is currently in use as a standard practice in emergency departments for managing mild and moderate hyperkalemia. This dosing regimen aligns with established clinical guidelines and is widely accepted as an effective approach in controlling potassium levels.
  Arms: Conventional Dose Therapy

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of a lower dose insulin compared to the conventional dose for treating mild to moderate hyperkalemia, a condition characterized by elevated serum potassium levels below 6.4 mmol/L. The study focuses on adult patients in the emergency department.

The primary objective is to determine whether the efficacy of lower doses of insulin and dextrose is non-inferior to conventional doses in reducing serum potassium levels in patients with mild to moderate hyperkalemia.

The research compares two regimens: 5 units of insulin with 25 mL of dextrose 50% versus 10 units of insulin with 50 mL of dextrose 50%, assessing the mean reduction in serum potassium levels, the incidence of hypoglycemia, and the risk of extravasation injury.

Participants will be monitored in the emergency department for 6 hours. Serum potassium levels will be measured at 1, 2, 4, and 6 hours post-intervention, while blood glucose levels will be monitored at 30, 60, 90, 120, 240, 300, and 360 minutes post-intervention.

DETAILED DESCRIPTION:
The primary research question that guided the design of this study arose from the consideration of optimizing insulin and dextrose dosing in the management of mild to moderate hyperkalaemia, specifically in patients with serum potassium levels below 6.4 mmol/L. This focus acknowledges that severe hyperkalaemia necessitates higher insulin doses, often accompanied by a corresponding increase in dextrose, to achieve a rapid and significant reduction in serum potassium levels. However, the necessity of administering the full conventional dose of insulin and dextrose in moderate hyperkalaemia is still unclear. Investigators hypothesize that a lower dose regimen may achieve similar efficacy in reducing serum potassium levels while potentially minimizing the risks associated with higher doses, such as hypoglycaemia and extravasation injury.

Previous studies have reported reductions in potassium ranging from 0.6-1.17 mmol/L following administration of lower dose of insulin. In this study, investigators aim to assess whether lower doses of insulin and dextrose are non-inferior to the standard dosing regimen. The non-inferiority margin has been defined as a reduction in serum potassium by 0.5 mmol/L for both treatment groups. This margin was carefully selected because a 0.5 mmol/L decrease in potassium is clinically significant, shifting the condition from moderate to mild hyperkalaemia, thereby reducing the risk of life-threatening arrhythmias. This threshold prioritises patient safety while potentially minimising adverse events, particularly hypoglycaemia, commonly linked to higher insulin doses.

Furthermore, if the lower doses are shown to be non-inferior, adverse events such as hypoglycaemia and extravasation could be reduced, enhancing the safety profile of hyperkalaemia management. This improvement represents a key secondary objective of the study and underscores the broader potential of dose optimisation.

Research specifically addressing optimal insulin dosing for hyperkalaemia is limited. Given limited research on optimal insulin dosing for hyperkalaemia, these findings could inform clinical guidelines, encouraging flexible, evidence-based dosing strategies in emergency and critical care settings

To determine the required sample size for this non-inferiority study comparing insulin dosages for treating moderate hyperkalaemia in the emergency department, investigators utilized a sample size calculation based on the method by Julious, 2004 and the following parameters.

Investigators aimed to detect whether the mean difference between the standard treatment and the experimental treatment does not exceed the non-inferiority limit of 0.5 mmol/L, with 80% power and a significance level of 0.05 for a two-sided test. Estimating a standard deviation of 0.68 mmol/L based on prior studies, and using the formula for comparing two means, 23 participants per arm are needed.

Including a 10% dropout rate, the total sample size required for the study is 50 participants, with 25 allocated to each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient >18 years old in emergency department (ED) with serum potassium 5.7 mmol/L to 6.4 mmol/L for non-haemolysed serum sample

Exclusion Criteria:

* Adolescent/ paediatric age group
* Patients who are in diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS)
* Pre-treatment blood glucose less than 4 mmol/L
* Requiring intraveneous (IV) infusion of insulin, nebulised salbutamol and IV sodium bicarbonate during screening
* Patient requiring resuscitation (ie: hemodynamically unstable) or requiring high flow oxygen (face mask > 5L/min) or Modified Early Warning Score > 4 during recruitment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean potassium difference between baseline and 1 hour post therapy | From administration of actrapid to the first hour after administration of actrapid
  The difference in serum potassium level between baseline and one hour post therapy will be compared between the two arms

SECONDARY OUTCOMES:
Incidence of hypoglycaemia within 6 hours of insulin administration | From administration of actrapid until the 6 hours after administration of actrapid
  Bedside glucose levels will be measured at 30, 60, 90, 120, 240, 300, and 360 minutes after insulin administration. Episodes of hypoglycemia (< 4.0 mmol/L) will be recorded.
Number of patients requiring rescue treatment for persistent hyperkalaemia (> 5.7 mmol/L) despite initial treatment | From administration of actrapid until the 6 hours after administration of actrapid
  Patients requiring rescue treatment for hyperkalemia, in both arms, will be documented and analyzed in this study
Mortality in patients within 7 days | From enrolment to 7 days after receiving interventional treatment
  Any reported mortality within 7 days as documented in the Electronic Medical Records, will be recorded and analyzed in the study.

CONTACTS AND LOCATIONS:
Overall Officials: NURUL ELLMY ABDUL RAZAK, MBBCh, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) will be shared. This includes de-identified participant data, study protocol, and statistical analysis plan. Data will be shared with researchers upon request and approval of a study proposal. Sharing will occur after publication of the trial results and will be made available via a secure data repository.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: De-identified Individual Participant Data (IPD), including demographic data, serum potassium levels, blood glucose levels, and treatment outcomes, will be shared with qualified researchers who submit a scientifically sound proposal. Researchers must provide detailed objectives, planned analyses, and compliance with ethical and privacy standards.
  Study Protocol and Informed Consent Form (ICF) will be available upon request. Proposals should be submitted via email to the Principal Investigator.

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group. KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney Int. 2024 Apr;105(4S):S117-S314. doi: 10.1016/j.kint.2023.10.018. No abstract available. PMID 38490803
- [Background] Verdier M, DeMott JM, Peksa GD. A comparison of insulin doses for treatment of hyperkalaemia in intensive care unit patients with renal insufficiency. Aust Crit Care. 2022 May;35(3):258-263. doi: 10.1016/j.aucc.2021.05.004. Epub 2021 Jun 21. PMID 34167889
- [Background] Schafers S, Naunheim R, Vijayan A, Tobin G. Incidence of hypoglycemia following insulin-based acute stabilization of hyperkalemia treatment. J Hosp Med. 2012 Mar;7(3):239-42. doi: 10.1002/jhm.977. PMID 22489323
- [Background] Pierce DA, Russell G, Pirkle JL Jr. Incidence of Hypoglycemia in Patients With Low eGFR Treated With Insulin and Dextrose for Hyperkalemia. Ann Pharmacother. 2015 Dec;49(12):1322-6. doi: 10.1177/1060028015607559. Epub 2015 Sep 28. PMID 26416951
- [Background] Pearson SC, O'Connor K, Keller K, Hodge TJ, Nesbit R. Efficacy of standard- vs reduced-dose insulin for treatment of hyperkalemia: A quasi-experiment. Am J Health Syst Pharm. 2022 Feb 18;79(Suppl 1):S13-S20. doi: 10.1093/ajhp/zxab382. PMID 34597356
- [Background] Moussavi K, Nguyen LT, Hua H, Fitter S. Comparison of IV Insulin Dosing Strategies for Hyperkalemia in the Emergency Department. Crit Care Explor. 2020 Apr 29;2(4):e0092. doi: 10.1097/CCE.0000000000000092. eCollection 2020 Apr. PMID 32426734
- [Background] LaRue HA, Peksa GD, Shah SC. A Comparison of Insulin Doses for the Treatment of Hyperkalemia in Patients with Renal Insufficiency. Pharmacotherapy. 2017 Dec;37(12):1516-1522. doi: 10.1002/phar.2038. Epub 2017 Nov 27. PMID 28976587
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Humphrey TJL, James G, Wilkinson IB, Hiemstra TF. Clinical outcomes associated with the emergency treatment of hyperkalaemia with intravenous insulin-dextrose. Eur J Intern Med. 2022 Jan;95:87-92. doi: 10.1016/j.ejim.2021.09.018. Epub 2021 Oct 5. PMID 34625340
- [Background] Garcia J, Pintens M, Morris A, Takamoto P, Baumgartner L, Tasaka CL. Reduced Versus Conventional Dose Insulin for Hyperkalemia Treatment. J Pharm Pract. 2020 Jun;33(3):262-266. doi: 10.1177/0897190018799220. Epub 2018 Sep 6. PMID 30189765
- [Background] Finder SN, McLaughlin LB, Dillon RC. 5 versus 10 Units of Intravenous Insulin for Hyperkalemia in Patients With Moderate Renal Dysfunction. J Emerg Med. 2022 Mar;62(3):298-305. doi: 10.1016/j.jemermed.2021.10.027. Epub 2022 Jan 17. PMID 35058093
- [Background] Chothia MY, Humphrey T, Schoonees A, Chikte UME, Davids MR. Hypoglycaemia due to insulin therapy for the management of hyperkalaemia in hospitalised adults: A scoping review. PLoS One. 2022 May 12;17(5):e0268395. doi: 10.1371/journal.pone.0268395. eCollection 2022. PMID 35552566
- See also: UKKA Clinical Practice Guideline - Management of Hyperkalaemia in Adults - October 2023 — https://www.ukkidney.org/sites/default/files/FINAL%20VERSION%20-%20UKKA%20CLINICAL%20PRACTICE%20GUIDELINE%20-%20MANAGEMENT%20OF%20HYPERKALAEMIA%20IN%20ADULTS%20-%20191223_0.pdf